CLINICAL TRIAL: NCT01045941
Title: Phase II Study of Adjuvant Gemcitabine Started One Week After Laparoscopic
Brief Title: Safety Study of Adjuvant Gemcitabine Started One Week After Laparoscopic Distal Pancreatectomy for Adenocarcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was never initiated
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00031399
Record Dates: First submitted 2009-12-09; First posted 2010-01-11 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Pancreatic Neoplasms
Keywords: Distal Pancreas; Adenocarcinoma; Laparoscopic; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with distal pancreatic cancer (Experimental): Patients with distal pancreatic cancer amenable to a laparoscopic distal pancreatectomy
  Interventions: Drug: Gemcitabine/Gemzar; Procedure: Laparoscopic Distal pancreatectomy

INTERVENTIONS:
Drug: Gemcitabine/Gemzar — Six cycles of Gemcitabine will be given. Each cycle of Gemcitabine comprises of Gemcitabine 1000 mg/m2 as a 30 minute infusion once weekly for 3 weeks with a fourth week off.
Procedure: Laparoscopic Distal pancreatectomy — Laparoscopic resection of the distal pancreas

SUMMARY:
We believe that laparoscopic distal pancreatectomy for cancer allows quicker recovery and significantly reduces the chances of postoperative wound breakdown. This will shorten the wait time required to begin adjuvant therapy to one week after surgery thereby combating the micrometastasis unseen at the time of surgery. Prognosis for patients with pancreatic cancer will therefore improve along with decreasing the incidence of locoregional recurrence.

DETAILED DESCRIPTION:
Gemcitabine-based chemo¬therapy remains the cornerstone for treatment of locally advanced or metastatic pancreatic cancer. Other novel chemotherapeutic combinations have been investigated in clinical trials, but the overall conclusions are that these agents have failed to improve outcomes. Our hypothesis is that nodal and hematologic micrometastasis make pancreas cancer a systemic problem at the time of surgery. Waiting the traditional six weeks to begin adjuvant therapy allows this very aggressive cancer to metastasize while the patient is waiting to begin therapy. This leads to the increased incidence of locoregional recurrence and poor prognosis. We believe that laparoscopic distal pancreatectomy for cancer allows quicker recovery and significantly reduces the chances of postoperative wound breakdown. This will shorten the wait time required to begin adjuvant therapy to one week after surgery thereby combating the micrometastasis unseen at the time of surgery. Prognosis for patients with pancreatic cancer will therefore improve along with decreasing the incidence of locoregional recurrence.

Methods: We will perform a prospective, non-randomized phase II study with patients undergoing laparoscopic distal pancreatectomy for pancreatic adenocarcinoma at Johns Hopkins Hospital. Gemcitabine will be given as a single-agent chemotherapy regimen one week following laparoscopic distal pancreatectomy according to the protocol designed by our medical oncologist. Six cycles of gemcitabine will be given. The patients will be followed in the medical oncology clinic weekly. Our Primary outcome variable will be all cause postoperative morbidity. Our sample size will be small (6-10 patients) as this is a Phase II study. Early termination rules include development of prohibitive toxicity or death. Our endpoints are an improvement in overall survival, quality of life, progression free survival, or disease free survival. Exclusion criteria will include patients with T4 or M1 disease, R2 resection margin, preoperative therapy, or if adjuvant therapy status was unknown.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients older than 18 with clinical diagnosis of distal pancreas adenocarcinoma

Exclusion Criteria:

* Patients with T4 or M1 disease, R2 resection margin, preoperative therapy, or if adjuvant therapy status was unknown.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To determine if it is safe to administer gemcitabine to patients with pancreatic cancer one week after laparoscopic distal pancreatectomy. | 1 year

SECONDARY OUTCOMES:
To determine the if the 1-year survival in patients with pancreatic cancer is improved with administration of gemcitabine one week following laparoscopic distal pancreatectomy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Makary, MD, MPH, Principal Investigator — Johns Hopkins University Department of Surgery
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Crane CH, Abbruzzese JL, Evans DB, Wolff RA, Ballo MT, Delclos M, Milas L, Mason K, Charnsangavej C, Pisters PW, Lee JE, Lenzi R, Vauthey JN, Wong AB, Phan T, Nguyen Q, Janjan NA. Is the therapeutic index better with gemcitabine-based chemoradiation than with 5-fluorouracil-based chemoradiation in locally advanced pancreatic cancer? Int J Radiat Oncol Biol Phys. 2002 Apr 1;52(5):1293-302. doi: 10.1016/s0360-3016(01)02740-7. PMID 11955742
- [Background] Kachnic LA, Shaw JE, Manning MA, Lauve AD, Neifeld JP. Gemcitabine following radiotherapy with concurrent 5-fluorouracil for nonmetastatic adenocarcinoma of the pancreas. Int J Cancer. 2001 Apr 20;96(2):132-9. doi: 10.1002/ijc.1008. PMID 11291097
- [Background] Regine WF, Winter KA, Abrams RA, Safran H, Hoffman JP, Konski A, Benson AB, Macdonald JS, Kudrimoti MR, Fromm ML, Haddock MG, Schaefer P, Willett CG, Rich TA. Fluorouracil vs gemcitabine chemotherapy before and after fluorouracil-based chemoradiation following resection of pancreatic adenocarcinoma: a randomized controlled trial. JAMA. 2008 Mar 5;299(9):1019-26. doi: 10.1001/jama.299.9.1019. PMID 18319412